CLINICAL TRIAL: NCT01494675
Title: Clinical Impact of Procalcitonin to Shorten Antimicrobial Therapy in Septic Patients With Proven Bacterial Infection in an Intensive Care Setting
Brief Title: Procalcitonin as a Tool to Shorten Antibiotic Therapy in the ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Rodrigo Octavio Deliberato, ICU staff physician at Hospital Israelita Albert Einstein, Hospital Israelita Albert Einstein
Model: Parallel | Masking: Triple
Other Study IDs: PCT
Record Dates: First submitted 2011-12-13; First posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Sepsis
Keywords: procalcitonin; duration of the antibiotic therapy; sepsis
MeSH Terms: conditions — Sepsis | interventions — Procalcitonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: procalcitonin measurement — The patients assigned to the procalcitonin group had procalcitonin and C reactive protein levels measured at day 0 (bacteremia), 5 or 7 (if positive blood culture) and then every 48 hours until hosptital discharge, death or until the antibiotics were stopped. A predefined procalcitonin protocol was used together with the clinical outcome, to guide the physician´s decision to discontinue antibiotics.
  The procalcitonin protocol encouraged the physician to discontinue the antibiotics when: 1)procalcitonin dropped more than 90% from the baseline peak level or 2)an absolute value below 0,5ng/mL was reached. Cases in which the antibiotic treatment was continued against what the PCT values indicated were categorized as " antibiotic discontinuation overruling"

SUMMARY:
Recently, biomarkers like procalcitonin have been studied in order to help physicians to decrease the duration of the antibiotic therapy. The investigators objective was to assess whether the decrease in procalcitonin levels could be used to reduce the antibiotic therapy in critically ill patients with a proven infection without risking a worse outcome.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted in the intensive care unit with sepsis, severe sepsis and septic shock with a microbiologically confirmed infection (blood, urine, tracheal aspirate or bronchoalveolar fluid culture)

Exclusion Criteria:

* onset of the antibiotic therapy more than 48 hours before the date when the cultures were performed
* patients less than 18 years old
* known pregnancy
* infections requiring prolonged antibotic therapy such as endocarditis, hepatic or brain abscess, deep abscess, mediastinitis and osteomyelitis
* severe infection caused by virus, parasites, fungi or chronic prostatitis
* negative cultures in patients with suspected sepsis, severe sepsis or septic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
reducing the duration of antibiotic therapy | 2 years
  the primary objective was to assess if a procalcitonin measurement protocol can reduce the duration of antibiotic therapy in critically ill patients with sepsis, severe sepsis and septic shock with documented infection

SECONDARY OUTCOMES:
all cause mortality | 2 years
  The secondary endpoints were in-hospital mortality, ICU mortality, ICU length of stay, recurrence of the initial infection, analyis of the C-reative protein levels along with the procalcitonin protocol and costs

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo O Deliberato, M.D., Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Sâo Paulo, Brazil